CLINICAL TRIAL: NCT03482193
Title: The Association of Adolescents' Interactive and Critical Health Literacy With Their Overweight: a Study in a Medium Urban City in Belgium
Brief Title: Health Literacy and Overweight in Adolescents
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Isabelle Bragard, Professor, University of Liege
Other Study IDs: HL-ado-obésité
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents: Adolescents in 2nd or 4th year in secondary school, from 9 different schools in Liège, Belgium.

SUMMARY:
Obesity in children and adolescents has become a major public health problem in recent years. In Belgium, 20% of people aged between 2 and 17 are overweight and 7% suffer from obesity. While studies often associate this overweight with socio-economic level, other factors, such as health literacy (HL), may also play a role. Among adolescents, some studies have shown an association between the level of HL and the Body Mass Index (BMI). Our study aims to investigate the association between HL of adolescents and their BMI.

This is a cross-sectional survey among 9 high schools in a medium city of Belgium, including 254 high school students aged between 12-17 years. Health literacy was assessed by the Health Literacy Measure for Adolescents (HELMA). Student's age, sex, weight, size and parental socio-economic status are gathered in the medical file during the medical examination organized by the schools after obtaining the informed consent of the students and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Studying in one of the participating school
* Being in 2nd or 4th year
* Parental consent to participate

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents studying in 2nd or 4th year in one of the participating secondary school. Students in those years receive a medical examination, which facilitate the collect of data and made us chose to limit the participation to these 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Health Literacy | 1 day (At the inclusion in the study)
  The degree to which individuals can obtain, process and understand basic health information and services needed to make appropriate health decisions. It also includes the cognitive and social skills which determine the motivation and ability of individuals to gain access to, understand and use information in ways which promote and maintain good health. It is measured by the Health Literacy Measure for Adolescents (HELMA) (Ghanbari et al., 2016), which is composed of 44 items. Health literacy was categorized into 4 categories based on the score to the questionnaire: excellent, sufficient, problematic and inadequate.
Body Mass Index | 1 day (At the inclusion in the study)
  Calculated with the standard formula (weight/height²) and categorized into 4 categories (underweight, normal, overweight, obesity) according to the PNNS and IOTF-25 and -30 curves.
Parents' socio-economic status | 1 day (At the inclusion in the study)
  We collected the profession of the parents' through the adolescent's medical file, and categorized them into 4 categories: worker, employee, independent, unemployed.

SECONDARY OUTCOMES:
Language spoken at home | 1 day (At the inclusion in the study)
  Collected through a socio-demographic questionnaire
Education type | 1 day (At the inclusion in the study)
  General eduction versus other (differentiated, professional, transition, qualification). Collected through a socio-demographic questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Bragard, Study Director — Université de Liège
Locations (1):
- University of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided